CLINICAL TRIAL: NCT00936078
Title: The Living Kidney Donor Safety Study (Long-term Effects of Becoming a Living Kidney Donor)
Brief Title: The Living Kidney Donor Safety Study
Acronym: LKD
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Astellas Pharma Canada, Inc. (Industry); Novartis (Industry)
Responsible Party: Principal Investigator, Amit Garg, Associate Dean (Clinical Research - Schulich School of Medicine and Dentistry); Professor (Medicine - Western University); Nephrologist (London Health Sciences Centre); Director (ICES Western Facilitly) (As of October 19 2022), London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Other Study IDs: R-09-117; 6056 (15974E) (Other: REB)
Record Dates: First submitted 2009-07-07; First posted 2009-07-09 (Estimated); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Living Kidney Donation
Keywords: blood pressure; glomerular filtration rate; hypertension; kidney transplantation; living kidney donation; unilateral nephrectomy
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum Urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Non-donors/controls: Healthy normotensive people who have not donated a kidney including relatives or friends of the donor, or candidates who were ineligible to donate due to blood group or cross-match incompatibility. These non-donor/controls must meet all screening criteria (same as standard criteria donors).
- Living Kidney Donors: Living kidney donors who went on to donate their kidney. All donors were recruited and are divided into 2 groups:
  1. Standard criteria donors (meet all screening criteria)
  2. Expanded-criteria donors (did not meet one or more of the screening criteria)
  Expanded criteria donors will be examined in a separate protocol and analysis.

SUMMARY:
The main goal of this study is to understand the long-term effects of kidney donation on blood pressure, kidney function, and patient-reported health-related quality of life. Living kidney donors and non-donor controls will be studied before and after the living donor transplant. The donors and non-donors will be followed for a minimum of 5 years and a maximum of 15 years. Both groups will be made up of healthy normotensive adults. The purpose of this study is to see if there are any long-term differences between the two groups regarding:

1. risk of hypertension
2. rate of kidney decline
3. risk of albuminuria
4. changes in health-related quality of life

The study also looks to assess other outcomes, including:

1. understand and quantify the expenses incurred by donors
2. understand donor factors which influence recipient outcomes

The pilot version of this study (The Long Term Medical and Psychological Implications of Becoming a Living Kidney Donor: A Prospective Pilot Study) began in 2004. Donors and controls in the pilot study were given the opportunity to continue on in the main study once it started in 2009.

DETAILED DESCRIPTION:
Transplantation is the preferred treatment option for patients with kidney failure. Compared to dialysis, patients who receive a transplant have a substantial reduction in the risk of death, an improved quality of life, and decreased health care costs. The demand for kidneys has resulted in long waiting lists for deceased donor kidneys. Therefore, living kidney donations have been on the increase over the years in order to meet this demand for kidneys. Living donation also has the added benefit of a shorter waiting time, increased graft success and increased recipient survival compared to deceased donor transplantation.

Aside from the advantages for the recipient, living transplantation is a complex medical practice which we must conduct in a safe and ethical manner. The premise for accepting living donors is that the "minimal" risk of short and long-term medical harm realized by the donor is outweighed by the definite advantages to the recipient and potential psychosocial benefits of altruism to the donor. The short-term potential medical consequences for living kidney donors have been well established. Yet, the long-term implications of living kidney donation are far less certain. Potential medical risks include hypertension, reduced kidney function, albuminuria, premature cardiovascular disease, and death. Estimates of these outcomes vary substantially in the literature. As well, the potential long-term medical risks are also communicated inconsistently across transplant communities. It is accepted that most living donors experience increased self-esteem, feelings of well-being and an improved quality of life after their altruistic act. However, some donors have negative psychosocial outcomes which require further clarification. There is also a financial burden to the donor from the donation process. Concerns about future life, disability, and medical insurance have been raised. These issues will be addressed through this research study on the long term implications of donation. A better understanding of post-donation risk and the timing of new disease onset is critical for donor selection, informed consent, and follow-up. The study will assess the attributable risk of living kidney donation using study techniques that meet modern criteria for high methodological quality. Non-donors will have similar indicators of baseline health as donors and will complete the same schedule of follow-up assessments.

Data was collected as follows:

1. Pre-donation/baseline (informed consent was obtained, eligibility was assessed, surveys were completed, a basic physical exam was completed, blood and urine samples were collected and training on the home blood pressure machine was completed). This occurred for both donors and non-donor controls either on site or long distance.
2. Three months post-donation (mailed 3 month surveys)
3. Annual post-donation follow-up visits (mailed surveys and blood pressure machine, lab testing completed). The number of annual follow-up visits varied depending on the year of nephrectomy, or simulated nephrectomy year for controls (between 5 years to 15 years)

Living kidney donation is practiced with the expectation that minimal risks of donor harm are outweighed by psychological benefits of altruism to the donor and improved recipient health. Our multicentre prospective cohort study of living kidney donors will inform the practice and safety of living kidney donation, including transplant center medical policies on donor selection, patient counseling, informed consent, and long-term patient follow-up and care.

ELIGIBILITY:
Inclusion Criteria:

* Be able to speak and read English and/or French, and
* Be able to provide informed consent, and

AND

Subjects must either:

* Be approved by the LHSC team (or applicable medical team at the participating sites) as eligible to donate their kidney and donated a kidney,

OR

* Meet study eligibility for controls (non-donors) as follows:

Be between the ages of 18 and 70 years

Meet blood pressure criteria as follows:

* Blood pressure <140 mmHg systolic and <90 mmHg diastolic based on an average of at least 3 blood pressure measurements taken during the recruitment interview, or an average blood pressure < 140 mmHg systolic and < 90 mmHg diastolic based on a minimum of 12 readings taken at home.
* All participants need to successfully record at least 12 home blood pressure readings using the self-monitoring device to be eligible

Meet local lab criteria as follows:

* Documented pre-donation serum creatinine <115 µmol/L in men or <90 µmol/L in women, or Cockcroft-Gault estimated glomerular filtration rate >80 mL/min
* Urine dipstick test for protein is negative or if trace or 0.3 g/L, a random urine albumin to creatinine ratio <8 mg/mmol (70 mg/g)
* Urine dipstick test for hematuria is negative. Those with non-persistent hematuria are eligible to participate. Those with initial evidence of dipstick hematuria may have a second assessment. Test should not occur during menses. Test should be repeated if there is evidence of urinary tract infection once treated.
* Have a body mass index of <35 kg/m2

Exclusion Criteria:

* Be involved in another clinical study that would affect the outcome of this study.

AND

Control (non-donor) subjects must not:

* Ever have received dialysis, even for a short period of time
* Ever have had a kidney transplant
* Be taking any hypertension class medication for any reason
* Have any history of hypertension, currently or in the past
* Have plasma glucose of >7 mmol/L after a 6 hour fast (if available), or a two hour oral glucose test of >11.1 mmol/L (if available), or have a history of diabetes during pregnancy
* Have been symptomatic or had evidence of kidney stones any time in the past 3 years
* Have a known contraindication to anesthesia or surgery
* Be currently pregnant or have been pregnant in the past month
* Have a medical condition that would prevent him or her from becoming a kidney donor (e.g. history of renal disease, permanent protein in urine, cancer other than cured non-melanoma skin cancer, cardiovascular disease, pulmonary disease, diabetes)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The donors will come from the identified population of people who will be donating their kidney at the hospital sites participating in this study.
  The non-donor population will be people who the donors identify and ask to act as their control person. As well, controls will also be found using pamphlet and poster board advertising.
Sampling Method: Non-Probability Sample
Enrollment: 1438 (Actual)
Dates: Start 2009-09 (Actual); Primary Completion 2021-11 (Actual); Study Completion 2022-03 (Actual)

PRIMARY OUTCOMES:
Hypertension | Annually (one data collection per year) for a minimum of 5 years to a maximum of 15 years after donation (baseline)
  Incident hypertension will be adjudicated by a physician who is blinded to the participant's donation status. Adjudication will occur if a participant meets the following criteria in follow-up: (1) the participant reports a physician diagnosis of hypertension, (2) the participant reports taking medication for hypertension, or (3) the participant has a systolic blood pressure (SBP) ≥140 or a diastolic blood pressure (DBP) ≥90 mmHg based on the average blood pressure (BP) measurements at any follow-up visit. Stage 1 hypertension will be defined as SBP/DBP 130 to 139/80 to 89 mmHg. We will also assess the average change in SBP and DBP over time accounting for the use of antihypertensive medications. Donors with pre-donation hypertension will be excluded from this primary analysis.

SECONDARY OUTCOMES:
Kidney Function | Annually (one data collection per year) for a minimum of 5 years to a maximum of 15 years after donation (baseline)
  We will assess the annualized change in eGFR over time (in mL/min per 1.73 m2 per year) in donors and non-donors using all available eGFR measurements, setting the starting eGFR value to be the one obtained (1) 1 year after the nephrectomy date (or 1 year after the assigned nephrectomy date for non-donors), (2) 3 years after the nephrectomy date, and (3) at baseline (pre-donation). We will also examine the proportion of participants whose eGFR fell below 60 mL/min per 1.73 m2 in follow-up, the proportion whose eGFR fell below 45 mL/min per 1.73 m2, and the proportion whose eGFR fell below 30 mL/min per 1.73 m2.
Albuminuria | Annually (one data collection per year) for a minimum of 5 years to a maximum of 15 years after donation (baseline)
  We will compare the geometric mean albumin-to-creatinine ratio in donors versus non-donors at the final follow-up visit, adjusted for the baseline (pre-donation) value. Values that are too low to measure will be recoded as 0.2 mg/mmol. We will also examine the proportion of participants who have an albumin-to-creatinine ratio ≥3 mg/mmol (≥30 mg/g) or >30 mg/mmol (>300 mg/g) at any time in follow-up.
Hypertension, an eGFR<60, and/or albuminuria | Annually (one data collection per year) for a minimum of 5 years to a maximum of 15 years after donation (baseline)
  We will examine the proportion of participants who develop hypertension, an eGFR <60 mL/min per 1.73 m2, or an albumin-to-creatinine ratio ≥3 mg/mmol. This outcome will be assessed as a composite, with death (expected to be rare during the follow-up period) treated as a competing event. We will also report the proportions of participants who develop (1) 2 or 3 of these components and (2) all 3 of these components.

OTHER OUTCOMES:
Death, kidney failure, and major cardiovascular events | Annually (one data collection per year) for a minimum of 5 years to a maximum of 15 years after donation (baseline)
  Death, kidney failure (i.e., a persistent eGFR less than 15 mL/min per 1.73 m2, receipt of dialysis for any duration, or receipt of a kidney transplant), and major cardiovascular events (i.e., myocardial infarction, stroke, or a cardiovascular procedure such as coronary angioplasty or coronary bypass surgery) will be assessed from the annual survey and from medical records, with adjudication conducted by a physician blinded to donation status. These outcomes will be assessed individually and as a composite.
Tinnitus (tracer outcome) | Annually (one data collection per year) for a minimum of 5 years to a maximum of 15 years after donation (baseline)
  Tinnitus (the perception of chronic ringing or noise in the ears) will be examined as a tracer outcome (i.e., a marker of self-report bias) because it is expected to be similar in donors and non-donors. Donors and non-donors with a history of tinnitus at enrollment will be excluded from this analysis.
Physical component summary (PCS) score of the 36-Item Short Form Survey (SF-36) | Annually (one data collection per year) for a maximum of 5 years, occurring up to a maximum of 15 years after donation (baseline)
  The PCS is derived from the following 8 domains of the SF-36 survey: physical functioning, role physical, bodily pain, general health perceptions, energy/vitality, social functioning, role emotional, and mental health. The PCS is scored according to documented procedures using Canadian or Australian normative data as appropriate, and ranges from 0 to 100 with higher scores representing better health status.
Mental component summary (MCS) score of the 36-Item Short Form Survey (SF-36) | Annually (one data collection per year) for a maximum of 5 years, occurring up to a maximum of 15 years after donation (baseline)
  The MCS is derived from the following 8 domains of the SF-36 survey: physical functioning, role physical, bodily pain, general health perceptions, energy/vitality, social functioning, role emotional, and mental health. The MCS is scored according to documented procedures using Canadian or Australian normative data as appropriate, and ranges from 0 to 100 with higher scores representing better health status."
Beck Depression Index (BDI) score | Annually (one data collection per year) for a maximum of 5 years, occurring up to a maximum of 15 years after donation (baseline)
  Depression will be assessed using the Beck Depression Inventory. The BDI has 21 items and assesses symptoms experienced over the past week. Scores range from 0 (no depression) to 63 (severe depression).
Beck Anxiety Inventory (BAI) score | Annually (one data collection per year) for a maximum of 5 years, occurring up to a maximum of 15 years after donation (baseline)
  Anxiety will be assessed using the Beck Anxiety Inventory. The BAI has 21 items and assesses symptoms experienced over the past month. Scores range from 0 (no anxiety) to 63 (severe anxiety).

CONTACTS AND LOCATIONS:
Overall Officials: Amit Garg, PhD, MD, Principal Investigator — London Health Sciences Centre
Locations (13):
- Sir Charles Gairdner Hospital, Perth, Australia
- Canada (12):
  - Foothills Medical Centre, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - St. Paul's Hospital, Vancouver, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - Health Sciences Centre, Winnipeg, Manitoba
  - Queen Elizabeth II Hospital, Halifax, Nova Scotia
  - St. Joseph's Hospital, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - The Montreal General Hospital, Montreal, Quebec

REFERENCES:
- [Background] Garg AX, Arnold JB, Cuerden M, Dipchand C, Feldman LS, Gill JS, Karpinski M, Klarenbach S, Knoll GA, Lok C, Miller M, Monroy-Cuadros M, Nguan C, Prasad GVR, Sontrop JM, Storsley L, Boudville N. The Living Kidney Donor Safety Study: Protocol of a Prospective Cohort Study. Can J Kidney Health Dis. 2022 Oct 28;9:20543581221129442. doi: 10.1177/20543581221129442. eCollection 2022. PMID 36325263
- [Result] Garcia-Ochoa C, Feldman LS, Nguan C, Monroy-Caudros M, Arnold JB, Barnieh L, Boudville N, Cuerden MS, Dipchand C, Gill JS, Karpinski M, Klarenbach S, Knoll G, Lok CE, Miller M, Prasad GVR, Sontrop JM, Storsley L, Garg AX. Impact of Perioperative Complications on Living Kidney Donor Health-Related Quality of Life and Mental Health: Results From a Prospective Cohort Study. Can J Kidney Health Dis. 2021 Aug 11;8:20543581211037429. doi: 10.1177/20543581211037429. eCollection 2021. PMID 34394947
- [Result] Habbous S, Arnold J, Begen MA, Boudville N, Cooper M, Dipchand C, Dixon SN, Feldman LS, Gozdzik D, Karpinski M, Klarenbach S, Knoll GA, Lam NN, Lentine KL, Lok C, McArthur E, McKenzie S, Miller M, Monroy-Cuadros M, Nguan C, Prasad GVR, Przech S, Sarma S, Segev DL, Storsley L, Garg AX; Donor Nephrectomy Outcomes Research (DONOR) Network. Duration of Living Kidney Transplant Donor Evaluations: Findings From 2 Multicenter Cohort Studies. Am J Kidney Dis. 2018 Oct;72(4):483-498. doi: 10.1053/j.ajkd.2018.01.036. Epub 2018 Mar 24. PMID 29580662
- [Result] Przech S, Garg AX, Arnold JB, Barnieh L, Cuerden MS, Dipchand C, Feldman L, Gill JS, Karpinski M, Knoll G, Lok C, Miller M, Monroy M, Nguan C, Prasad GVR, Sarma S, Sontrop JM, Storsley L, Klarenbach S; Donor Nephrectomy Outcomes Research (DONOR) Network. Financial Costs Incurred by Living Kidney Donors: A Prospective Cohort Study. J Am Soc Nephrol. 2018 Dec;29(12):2847-2857. doi: 10.1681/ASN.2018040398. Epub 2018 Nov 7. PMID 30404908
- [Result] Barnieh L, Klarenbach S, Arnold J, Cuerden M, Knoll G, Lok C, Sontrop JM, Miller M, Ramesh Prasad GV, Przech S, Garg AX; Donor Nephrectomy Outcomes Research (DONOR) Network. Nonreimbursed Costs Incurred by Living Kidney Donors: A Case Study From Ontario, Canada. Transplantation. 2019 Jun;103(6):e164-e171. doi: 10.1097/TP.0000000000002685. PMID 31246933
- [Result] Garcia-Ochoa C, Feldman LS, Nguan C, Monroy-Cuadros M, Arnold J, Boudville N, Cuerden M, Dipchand C, Eng M, Gill J, Gourlay W, Karpinski M, Klarenbach S, Knoll G, Lentine KL, Lok CE, Luke P, Prasad GVR, Sener A, Sontrop JM, Storsley L, Treleaven D, Garg AX; Donor Nephrectomy Outcomes Research (DONOR) Network. Perioperative Complications During Living Donor Nephrectomy: Results From a Multicenter Cohort Study. Can J Kidney Health Dis. 2019 Jul 18;6:2054358119857718. doi: 10.1177/2054358119857718. eCollection 2019. PMID 31367455
- [Result] Barnieh L, Arnold JB, Boudville N, Cuerden MS, Dew MA, Dipchand C, Feldman LS, Gill JS, Karpinski M, Klarenbach S, Knoll G, Lok C, Miller M, Monroy M, Nguan C, Prasad GVR, Sontrop JM, Storsley L, Garg AX; Donor Nephrectomy Outcomes Research (DONOR) Network. Living Kidney Donors' Financial Expenses and Mental Health. Transplantation. 2021 Jun 1;105(6):1356-1364. doi: 10.1097/TP.0000000000003401. PMID 33741846
- [Result] Barnieh L, Kanellis J, McDonald S, Arnold J, Sontrop JM, Cuerden M, Klarenbach S, Garg AX, Boudville N; Donor Nephrectomy Outcomes Research (DONOR) Network. Direct and indirect costs incurred by Australian living kidney donors. Nephrology (Carlton). 2018 Dec;23(12):1145-1151. doi: 10.1111/nep.13205. PMID 29215180
- [Result] Garg AX, Arnold JB, Cuerden MS, Dipchand C, Feldman LS, Gill JS, Karpinski M, Klarenbach S, Knoll G, Lok CE, Miller M, Monroy-Cuadros M, Nguan C, Prasad GVR, Sontrop JM, Storsley L, Boudville N. Hypertension and Kidney Function After Living Kidney Donation. JAMA. 2024 Jul 23;332(4):287-299. doi: 10.1001/jama.2024.8523. PMID 38780499